CLINICAL TRIAL: NCT00721188
Title: Single-Dose Pharmacokinetics of Venofer (Iron Sucrose Injection) in Non-Dialysis Dependent (NDD-CKD) Pediatric Patients Receiving or Not Receiving Erythropoiesis Stimulating Agents (ESA's)
Brief Title: Iron Sucrose in Non-Dialysis Dependent (NDD-CKD) Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN05033
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated

ARMS (1):
- Pharmacokinetic Population (Experimental): All subjects who received study drug and completed Pharmacokinetic testing through 24 hours post-dose.
  Interventions: Drug: Venofer

INTERVENTIONS:
Drug: Venofer — Single dose of 7mg intravenous (IV) of iron per kg of body weight for a maximum of 200mg iron IV.

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics of Venofer (Iron Sucrose Injection) in NDD-CKD pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 12 to < or = 16 years
* Parent and/or legal guardian able to give informed consent
* Subject able to give written assent for participating in the study
* NDD-CKD defined as: kidney damage for 3 months or longer, or GFR < 60 for 3 months or longer
* Hemoglobin indicative of anemia
* Ferritin indicative of iron deficiency anemia
* If appropriate, subject must be willing to use an accepted form of birth control from time of screening through the follow-up period

Exclusion Criteria:

* Known history of hypersensitivity to any component of Venofer
* Parenteral iron within 14 days of the screening visit
* Dialysis dependent-CKD
* Chronic or serious active infection
* Pregnancy or lactation
* Subjects with causes of iron deficiency anemia other than CKD
* Blood transfusion within the last month or anticipated during the study
* Body weight < 55 pounds
* Received an investigational drug within 30 days before screening

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 2006 to July 2008 Location: Hospital
Groups:
- Venofer (Iron Sucrose Injection): All subjects who received study drug and completed Pharmacokinetic testing through 24 hours post-dose.
Period: Overall Study
Arm/Group | Venofer (Iron Sucrose Injection)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  Mexico | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 9
ug/dL | 8545.33 (4118.54)

2. Primary Outcome: Time to Maximum Serum Concentration (Tmax)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 9
hour | 0.56 (0.17)

3. Primary Outcome: Serum Terminal Phase Elimination Half-life (T1/2)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 8
hour | 8.04 (4.51)

4. Primary Outcome: Area Under the Serum Concentration-time Curve From Time of Dosing to the Last Quantifiable Measurable Serum Concentration (AUC 0-last)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: ug*hr/dL
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 9
ug*hr/dL | 31304.84 (9850.48)

5. Primary Outcome: Area Under the Serum Concentration-time Curve Extrapolated to Infinity (AUC 0-∞)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 8
ug/dL | 36293.39 (12228.76)

6. Primary Outcome: Terminal Phase Elimination Rate Constant (λz)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 8
1/hour | 0.15 (0.15)

7. Secondary Outcome: Total Body Clearance (Cl)
Description: Total body clearance: Cl = Dose/Area Under the Serum Concentration-time Curve Extrapolated to Infinity (AUC 0-∞)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours.
Measure: Mean (Standard Deviation); unit: dL/hour
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 8
dL/hour | 6.03 (1.81)

8. Secondary Outcome: Initial Volume of Distribution (Vdc)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: dL
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 9
dL | 22.46 (14.12)

9. Secondary Outcome: Volume of Distribution Based on the Terminal Phase (Vdarea)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: dL
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 8
dL | 63.83 (30.28)

10. Secondary Outcome: Volume of Distribution at Steady State (Vdss)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: dL
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 8
dL | 40.27 (20.00)

11. Secondary Outcome: Mean Residence Time (MRtime)
Time Frame: Pre-dose and post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, and 12 hours.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 8
hour | 7.16 (4.08)

12. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE's)
Time Frame: Day of initial treatment with Venofer through 30 days after study treatment
Measure: Number; unit: participants
Arm/Group | Venofer (Iron Sucrose Injection)
Number analyzed (Participants) | 11
participants | 0

ADVERSE EVENTS:
Time Frame: Day of initial treatment with Venofer through 30 days after study treatment
Arm/Group | Venofer (Iron Sucrose Injection)
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venofer (Iron Sucrose Injection) (N=11)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less